CLINICAL TRIAL: NCT00543270
Title: Endologix Powerlink Long-Term Follow-up Study
Brief Title: Powerlink Bifurcated Stent Graft Long-Term Follow-up Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endologix (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TP00-005/CP04-001
Record Dates: First submitted 2007-10-10; First posted 2007-10-12 (Estimated); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: EVAR; AAA; Aneurysm; Powerlink
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aneurysm | interventions — Conversion to Open Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Endovascular Repair - EVAR (Powerlink System) (Experimental): EVAR (Powerlink System)
  Interventions: Device: Powerlink infrarenal bifurcated stent graft delivery system
- Open Surgical Control (Active Comparator): Open Surgical Control
  Interventions: Procedure: Open Surgery

INTERVENTIONS:
Device: Powerlink infrarenal bifurcated stent graft delivery system — Endovascular abdominal aortic aneurysm repair
  Other Names: Powerlink Stent Graft Delivery System
  Arms: Endovascular Repair - EVAR (Powerlink System)
Procedure: Open Surgery — Open surgical abdominal aortic aneurysm repair
  Arms: Open Surgical Control

SUMMARY:
Endologix Infrarenal Bifurcated Stent Graft Study

ELIGIBILITY:
Inclusion Criteria:

* All surviving patients from the original study cohort who received the Powerlink device
* All surviving patients from the original study cohort who were assigned to the open surgical control arm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2005-10; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
No of Subjects with Major adverse events | At 1 Year
  Aneurysm-related mortality, aneurysm rupture, conversion to open repair, coronary intervention, myocardial infarction, renal failure, respiratory failure, secondary procedure, and stroke
All Cause Mortality | At 1 Year
  No of deaths reported through 1 year

SECONDARY OUTCOMES:
Stent Graft Performance | 30 Days
  Total number of Subjects with Stent fracture, Stent Graft Migration, Stent Graft patency and Device Migration
Stent Graft Performance | 6 Months
  Total number of Subjects with Stent fracture, Stent Graft Migration, Stent Graft patency and Device Migration
Stent Graft Performance | Year 1
  Total number of Subjects with Stent fracture, Stent Graft Migration, Stent Graft patency and Device Migration
Stent Graft Performance | Year 2
  Total number of Subjects with Stent fracture, Stent Graft Migration, Stent Graft patency and Device Migration
Stent Graft Performance | Year 3
  Total number of Subjects with Stent fracture, Stent Graft Migration, Stent Graft patency and Device Migration
Stent Graft Performance | Year 4
  Total number of Subjects with Stent fracture, Stent Graft Migration, Stent Graft patency and Device Migration
Stent Graft Performance | Year 5
  Total number of Subjects with Stent fracture, Stent Graft Migration, Stent Graft patency and Device Migration
Clinical Utility Outcomes | During the Procedure
  Estimated anesthesia time, fluoroscopy time, procedure time
Clinical Utility Outcomes | During the Procedure
  Estimated blood loss (ml) and contrast volume (ml). Estimated blood loss records the approximate amount of blood that the patient lost during the surgery (ml) and contract volume is the volume of the contrast (ml) calculated during the procedure.
Clinical Utility Outcomes | up to 1 week
  Estimated ICU time
Clinical Utility Outcomes | up to 1 week
  Estimated Hospitalization Time
Aneurysm Morphology | 6 Months
  Change in aneurysm sac diameter from first post-procedural CT scan (30 days) to 6 Months
Aneurysm Morphology | Year 1
  Change in aneurysm sac diameter from first post-procedural CT scan (30 days) to Year 1
Aneurysm Morphology | Year 2
  Change in aneurysm sac diameter from first post-procedural CT scan (30 days) to Year 2
Aneurysm Morphology | Year 3
  Change in aneurysm sac diameter from first post-procedural CT scan (30 days) to Year 3
Aneurysm Morphology | Year 4
  Change in aneurysm sac diameter from first post-procedural CT scan (30 days) to Year 4
Aneurysm Morphology | Year 5
  Change in aneurysm sac diameter from first post-procedural CT scan (30 days) to Year 5

CONTACTS AND LOCATIONS:
Overall Officials: Rodney White, MD, Principal Investigator — University of California, Los Angeles
Locations (14):
- United States (14):
  - Arizona Heart Institute, Phoenix, Arizona
  - Harbor-UCLA Medical Center, Torrance, California
  - University of Illinois School of Medicine, Peoria, Illinois
  - SIU School of Medicine, Springfield, Illinois
  - Mercy Hospital, Des Moines, Iowa
  - Mayo Clinic, Rochester, Minnesota
  - Barnes Jewish Hospital, St Louis, Missouri
  - Advanced Vascular Associates, Morristown, New Jersey
  - Cleveland Clinic, Cleveland, Ohio
  - Oklahoma Cardiovascular Research Group, Oklahoma City, Oklahoma
  - University Hospital of Pennsylvania, Philadelphia, Pennsylvania
  - Greenville Hospital System, Greenville, South Carolina
  - Heart Hospital of South Dakota, Sioux Falls, South Dakota
  - Vascular and Transplant Specialists, Norfolk, Virginia

REFERENCES:
- [Result] Carpenter JP. The Powerlink bifurcated system for endovascular aortic aneurysm repair: four-year results of the US multicenter trial. J Cardiovasc Surg (Torino). 2006 Jun;47(3):239-43. PMID 16760859
- [Result] Parmer SS, Carpenter JP; Endologix Investigators. Endovascular aneurysm repair with suprarenal vs infrarenal fixation: a study of renal effects. J Vasc Surg. 2006 Jan;43(1):19-25. doi: 10.1016/j.jvs.2005.09.025. PMID 16414382
- [Result] Wang GJ, Carpenter JP. EVAR in small versus large aneurysms: does size influence outcome? Vasc Endovascular Surg. 2009 Jun-Jul;43(3):244-51. doi: 10.1177/1538574408327570. Epub 2008 Dec 16. PMID 19088132
- [Result] Wang GJ, Carpenter JP; Endologix Investigators. The Powerlink system for endovascular abdominal aortic aneurysm repair: six-year results. J Vasc Surg. 2008 Sep;48(3):535-45. doi: 10.1016/j.jvs.2008.04.031. Epub 2008 Jul 16. PMID 18635335